CLINICAL TRIAL: NCT00017290
Title: A Phase III Trial To Evaluate The Safety And Efficacy Of Specific Immunotherapy, Recombinant Idiotype Conjugated To KLH With GM-CSF, Compared To Non-Specific Immunotherapy, KLH With GM-CSF, In Patients With Follicular Non-Hodgkin's Lymphoma
Brief Title: Combination Chemotherapy Followed By Vaccine Therapy Plus Sargramostim in Treating Patients With Stage III or Stage IV Non-Hodgkin's Lymphoma
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Genitope Corporation (Industry)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: CDR0000068673; GENITOPE-G2000-03; CUMC-0101-142; UCLA-0010061
Record Dates: First submitted 2001-06-06; First posted 2003-01-27 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2002-08

CONDITIONS: Lymphoma
Keywords: stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III grade 3 follicular lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; stage IV grade 3 follicular lymphoma
MeSH Terms: conditions — Lymphoma; Lymphoma, Follicular | interventions — keyhole-limpet hemocyanin; sargramostim; Cyclophosphamide; Prednisone; Vincristine

INTERVENTIONS:
Biological: autologous immunoglobulin idiotype-KLH conjugate vaccine
Biological: keyhole limpet hemocyanin
Biological: sargramostim
Drug: cyclophosphamide
Drug: prednisone
Drug: vincristine sulfate

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Vaccines may make the body build an immune response to kill cancer cells. It is not yet known which regimen of chemotherapy combined with vaccine therapy is more effective for non-Hodgkin's lymphoma.

PURPOSE: Randomized phase III trial to determine the effectiveness of combination chemotherapy followed by vaccine therapy plus sargramostim in treating patients who have stage III or stage IV non-Hodgkin's lymphoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the time to tumor progression in patients with stage III or IV follicular B-cell non-Hodgkin's lymphoma treated with cyclophosphamide, prednisone, and vincristine followed by immunotherapy with keyhole limpet hemocyanin with or without autologous tumor-derived immunoglobulin idiotype and adjuvant sargramostim (GM-CSF).
* Compare the efficacy of these immunotherapy regimens in terms of converting patients with partial response or unconfirmed complete response to clinical complete response.
* Compare the safety and toxic effects of these immunotherapy regimens in this patient population.
* Compare the time to treatment failure and survival of patients treated with these regimens.
* Correlate the induction of idiotype-specific immune response with clinical benefits of achieving molecular remission in these patients.
* Compare the quality of life of patients treated with these regimens.

OUTLINE: This is a randomized, double-blind, placebo-controlled, multicenter study.

Patients receive cyclophosphamide IV over 30-40 minutes and vincristine IV on day 1. Patients also receive oral prednisone on days 1-5. Treatment repeats every 21 days for 8 courses.

At 6 months after completion of chemotherapy, patients maintaining partial response (PR), complete response (CR), or unconfirmed complete response (CRU) receive immunotherapy. Patients are stratified according to participating center and baseline disease status (PR vs CR/CRU). Patients are randomized to one of two treatment arms.

* Arm I: Patients receive autologous tumor-derived immunoglobulin idiotype conjugated to keyhole limpet hemocyanin (KLH) subcutaneously (SC) on day 1 and adjuvant sargramostim (GM-CSF) SC on days 1-4 of weeks 0, 4, 8, 12, 16, 20, and 24.
* Arm II: Patients receive KLH alone SC on day 1 and GM-CSF SC on days 1-4 of weeks 0, 4, 8, 12, 16, 20, and 24.

Quality of life is assessed prior to first immunization, at 2-8 weeks after completion of immunizations, and then every 6 months for 30 months.

Patients are followed every 3 months for 1 year and then every 6 months thereafter. Patients also enroll in a long-term follow-up study for an additional 5 years.

PROJECTED ACCRUAL: A total of 360 patients (240 in arm I and 120 in arm II) will be accrued from the 480 patients biopsied for this study within 15-18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed stage III or IV follicular B-cell non-Hodgkin's lymphoma
* At least 1 bidimensionally measurable lesion by radiography, in addition to lesion removed for biopsy
* No clinical evidence of CNS involvement

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* WBC greater than 1,500/mm^3
* Platelet count greater than 100,000/mm^3

Hepatic:

* Bilirubin less than 1.5 times upper limit of normal (ULN)
* Hepatitis B surface antigen negative
* Hepatitis C antibody negative

Renal:

* Creatinine less than 1.5 times ULN

Other:

* No other malignancy within the past 5 years except adequately treated basal or squamous cell skin cancer or carcinoma in situ of the cervix
* No history of autoimmune disease
* HIV negative
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior antibody therapy for lymphoma

Chemotherapy:

* No prior cytotoxic therapy for lymphoma

Endocrine therapy:

* No prior corticosteroids for lymphoma
* At least 12 months since prior corticosteroids or immunosuppressants for other conditions
* Prior transient corticosteroids (prior to CT imaging) or optical solutions allowed

Radiotherapy:

* Prior radiotherapy for lymphoma (no more than 2 sites of limited disease) allowed

Surgery:

* See Disease Characteristics

Other:

* No concurrent participation in other therapeutic clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-11

CONTACTS AND LOCATIONS:
Overall Officials: David Hinds, Study Chair — Genitope Corporation
Locations (24):
- United States (21):
  - SuperGen, Incorporated, Dublin, California
  - California Cancer Care, Inc., Greenbrae, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Stanford Cancer Center at Stanford University Medical Center, Stanford, California
  - Rocky Mountain Cancer Centers - Midtown, Denver, Colorado
  - Shands Cancer Center at the University of Florida Health Science Center, Gainesville, Florida
  - Mountain States Tumor Institute - Boise, Boise, Idaho
  - Rush Cancer Institute at Rush University Medical Center, Chicago, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Greenebaum Cancer Center at University of Maryland Medical Center, Baltimore, Maryland
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Veterans Affairs Medical Center - Ann Arbor, Ann Arbor, Michigan
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - UNMC Eppley Cancer Center at the University of Nebraska Medical Center, Omaha, Nebraska
  - Cancer Center at Hackensack University Medical Center, Hackensack, New Jersey
  - New York Weill Cornell Cancer Center at Cornell University, New York, New York
  - Arthur G. James Cancer Hospital - Ohio State University, Columbus, Ohio
  - Cancer Institute at Oregon Health and Science University, Portland, Oregon
  - Sarah Cannon Cancer Center at Centennial Medical Center, Nashville, Tennessee
- Canada (3):
  - Cross Cancer Institute, Edmonton, Alberta
  - British Columbia Cancer Agency, Vancouver, British Columbia
  - Toronto Sunnybrook Regional Cancer Centre, Toronto, Ontario

REFERENCES:
- [Derived] Levy R, Ganjoo KN, Leonard JP, Vose JM, Flinn IW, Ambinder RF, Connors JM, Berinstein NL, Belch AR, Bartlett NL, Nichols C, Emmanouilides CE, Timmerman JM, Gregory SA, Link BK, Inwards DJ, Freedman AS, Matous JV, Robertson MJ, Kunkel LA, Ingolia DE, Gentles AJ, Liu CL, Tibshirani R, Alizadeh AA, Denney DW Jr. Active idiotypic vaccination versus control immunotherapy for follicular lymphoma. J Clin Oncol. 2014 Jun 10;32(17):1797-803. doi: 10.1200/JCO.2012.43.9273. Epub 2014 May 5. PMID 24799467